CLINICAL TRIAL: NCT06629051
Title: A Multicenter, Placebo-controlled Clinical Study of Berberine Hydrochloride in Preventing Recurrence and Carcinogenesis After Endoscopic Removal of Colorectal Adenomas：6-year Retrospective Follow-up Data
Brief Title: 6-year Follow-up Data After the Berberine Intervention Trial
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Seventh Medical Center of PLA Army General Hospital (Other); Zhongshan Hospital Xiamen University (Other); Nanfang Hospital, Southern Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Tianjin Medical University General Hospital (Other); the Tenth People's Hospital affiliated to Tongji University (Unknown)
Responsible Party: Principal Investigator, Jing-yuan Fang, MD, Ph. D, Division of Gastroenterology & Hepatology, Renji Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: LY2024-232-A
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Adenoma; Colorectal Cancer Control and Prevention; Colorectal Polyps
Keywords: berberine; colorectal adenoma; colorectal cancer; long term chemoprevention; colorectal polyps
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- berberine: post-intervention of berberine
  Interventions: Drug: Berberine Hydrochloride
- placebo: post-intervention of placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berberine Hydrochloride — post-intervention of berberine
  Groups: berberine
Drug: Placebo — Looks the same as berberine
  Groups: placebo

SUMMARY:
Colorectal cancer (CRC) is a common malignancy of the digestive tract, which constitutes a major public health burden. Almost 90% of CRC cases progress from precursor adenomatous polyps through adenoma-carcinoma sequence. Endoscopic detection and removal of colorectal adenoma (CRA) could reduce the incidence and mortality risk of CRC, but the recurrence rate is still high. Therefore, chemoprevention is quite important, not only solve the urgent public health problem, but also be cost-effective.

In 2020, the investigators published a multicenter, randomized, double-blind, placebo-controlled clinical study (NCT02226185) in the Lancet Gastroenterology & Hepatology. The result concluded that oral BBR for 2 years significantly reduced recurrence after endoscopic removal of CRA (RR 0.77, 95%CI 0.66-0.91; p=0.001). BBR also has a significant preventive effect on all polypoid lesions, including adenomas and serrated lesions (adjusted RR 0.78, 95%CI 0.66-0.91; p=0.002) . Does BBR still have a long-term protective effect on the recurrence of CRA after discontinuation? That's what the investigators concerned.

The present study is performed to observe and compare retrospectively the recurrence rate of CRAs in patients of the original BBR RCT study (NCT02226185) within 6 years after discontinuation of medication, including the overall recurrence rate of traditional adenomas within the first year, 1-3 years, 3-6 years, and the entire follow-up period of 6 years. The aim is to evaluate the long-term efficacy of BBR in preventing recurrence and carcinogenesis after endoscopic resection of CRAs.

ELIGIBILITY:
Inclusion Criteria: participants who completed the previous berberine intervention study (NCT02226185) Exclusion Criteria: no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We included 895 participants who completed the previous berberine intervention study (NCT02226185), including 432 participants in the BBR group and 463 participants in the placebo group.
Sampling Method: Non-Probability Sample
Enrollment: 891 (Estimated)
Dates: Start 2024-10-04 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The recurrence rates of traditional colorectal adenomas within the follow-up period of 6 years | 6 years, 1-3 years, 3-6 years
  The cumulative recurrence rate of CRAs within the entire follow-up period of 6 years. The recurrence rates of CRAs within the first year, 1-3 years, 3-6 years. The number, size and location of all adenomas are assessed.

SECONDARY OUTCOMES:
The incidence rates of hyperplastic polyps and serrated adenomas within 6 years after discontinuation of medication | 6 years, 1-3 years, 3-6 years
  The recurrence rates within the first year, 1-3 years, 3-6 years, and the entire follow-up period of 6 years.
Subgroup analyses | 6 years, 1-3 years, 3-6 years
  For patients with advanced CRA or high-risk adenomas (including advanced CRA and multiple adenomas≥3），the recurrence rates of CRAs and polyps are further evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Yuan Fang, M.D, Ph.D, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
All included IPD
Supporting Information: Study Protocol, SAP